CLINICAL TRIAL: NCT00813436
Title: The Effect of Intranasal Administration of Oxytocin on Empathic Abilities of Healthy People and People Who Suffer From Schizophrenia.
Brief Title: The Effect of Intranasal Administration of Oxytocin on Empathic Abilities.
Acronym: 20070766
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Dr. Yechiel Levkovitz, Shalvata Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0007-07-SHA
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2008-12

CONDITIONS: Schizophrenia
Keywords: ToM; Theory of Mind; Simulation; Empathy; Oxytocin; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Oxytocin
  Interventions: Drug: Oxytocin (also: syntocinon, pitocin)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin (also: syntocinon, pitocin) — 24 IU for each subject (3 puffs in each nostril, 4 IU in each puff). each subject will receive a single administration, 40 minuets before task start time.
  Other Names: Novartis.
  Arms: 1
Drug: Placebo — saline liquid, intranasally administered
  Other Names: Weleda
  Arms: 2

SUMMARY:
Empathy constitutes one prominent ability of social cognition, which represents the human capability of understanding mental state of the other, and responding in sympathetic way. Two sets of theoretical mechanisms were designed in order to explain how empathy is possible. Theory of Mind (ToM)and Simulation.People who suffer from schizophrenia frequently exhibit social dysfunction, preventing them of a normal integration in healthy human environments. Recently it had been discovered that impairment in empathy and a specific impairment in effective TOM are mostly associated with the social malfunctioning of people who suffer from schizophrenia. One of the biological substances most connected to social cognition is the neuromodulator Oxytocin. Among its known involvement in uterine contractions and lactating females, numerous recent studies have found an indispensable role for Oxytocin in various complex prosocial behaviors such as maternal behavior, attachment, partner preference and trust. In the proposed study, we plan to examine the influence of a single dose of intranasal Oxytocin on the two primary mechanisms of empathy, namely mentalizing (Theory of Mind) and Simulation, both in healthy people and in people who suffer from schizophrenia.

DETAILED DESCRIPTION:
Social cognition encompasses a wide spectrum of abilities, enabling us to function properly in interpersonal interactions. Empathy constitutes one prominent ability of social cognition, which represents the human capability of understanding mental state of the other, and responding in sympathetic way (Leiberg & Anders, 2006). Two sets of theoretical mechanisms were designed in order to explain how empathy is possible. Theory of Mind (ToM) is usually regarded as a more cognitive mechanism of empathy, in which a theory we posses regarding the other enable us to infer his mental state. 'Simulation' processing is another different mechanism of empathy. In contrast to the ToM perspective, the simulation perspective asserts that understanding the other's state of mind is achieved by an inner representation of that mental state in our mind, thus simulating his mental state. Therefore, the simulation theory may be associated with more affective aspects of empathy.

Schizophrenia encompasses a wide spectrum of psychotic disorders, characterized by severe cognitive, emotional and behavioral impairments. People who suffer from schizophrenia frequently exhibit social dysfunction, preventing them of a normal integration in healthy human environments. Recently it had been discovered that impairment in empathy and a specific impairment in effective TOM are mostly associated with the social malfunctioning of people who suffer from schizophrenia.

One of the biological substances most connected to social cognition is the neuromodulator Oxytocin. Among its known involvement in uterine contractions and lactating females, numerous recent studies have found an indispensable role for Oxytocin in various complex prosocial behaviors such as maternal behavior, attachment, partner preference and trust. It was suggested that Oxytocin may mediate the beneficial affect of social support, and is found strongly involved in different kinds of attachment. In a recent study, Domes et al. (2006) found that an intranasal administration of a single dose of Oxytocin enhanced the ability to infer mental states as conveyed by the eyes region (RMET, Baron-Cohen et al. 1995). These findings suggest a mediating role for the ability to use social cues in order to infer the other mental states. In the proposed study, we plan to examine the influence of a single dose of intranasal Oxytocin on the two primary mechanisms of empathy, namely mentalizing (Theory of Mind) and Simulation, both in healthy people and in people who suffer from schizophrenia. Mentalizing will be assessed by a variation of a validated ToM task, which requires cognitive and affective mentalizing. Simulation will be tested in two different tasks: emotion recognition via a dynamic paradigm of facial expressions, and recognition of biological motion, which necessitates the identification of the emotion conveyed in a video clips of point light walkers. Both of these latter tasks have been associated with simulation processing.

ELIGIBILITY:
Inclusion Criteria (for schizophrenic patients):

1. Range of age between 18 and 45 years.
2. The patient is diagnosed as suffering from schizophrenia by 2 independent psychiatrists, according to DSM-IV criteria.
3. The participant is able to commit to 2 trials with 7 days interval.
4. The participant has been informed orally and in writing and has given his/her written consent.
5. When necessary, a psychiatrist has determined the patient's ability to agree, orally and in writing.

Inclusion Criteria (for healthy patients):

1. Range of age between 18 and 45 years.
2. The participant is able to commit to 2 trials with 7 days interval.
3. The participant has been informed orally and in writing and Has given his/her written consent.

Exclusion Criteria (for schizophrenic patients):

1. The participant is suffering from other acute, unstable, significant or untreated medical Illness, including arrhythmia and head injury.
2. The participant is suffers from an axis II disorder of DSM-IV.
3. The participant has history of alcohol or drug abuse.
4. The participant is pregnant or breast-feeding.
5. The participant suffers from mental retardation (IQ less than 75).
6. The participant has any disturbance in visuomotor coordination.
7. The participant has smoked a cigarette in the day of the trial.
8. High suicidal risk, as determined by the treating physician.

Exclusion Criteria (for healthy patients):

1. The participant is suffering from acute, unstable, significant or untreated medical Illness, including arrhythmia and head injury.
2. The participant has history of alcohol or drug abuse.
3. The participant is pregnant or breast-feeding.
4. The participant suffers from mental retardation (IQ less than 75).
5. The participant has any disturbance in visuomotor coordination.
6. The participant has smoked a cigarette in the day of the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
accuracy level (in percentage) and reaction time (in milliseconds) of emotional facial expressions recognition in a dynamic emotional facial expressions task. | end of second trial for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Levkovitz, MD, Principal Investigator — Shalvata Mental Health Center; Simone Shamay-Tsoory, MA, Study Director — University of Haifa
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel